CLINICAL TRIAL: NCT04196283
Title: A Phase 1b, Multicenter, Open-Label Study to Determine the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of ABBV-368 Plus Tilsotolimod and Other Therapy Combinations in Subjects With Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: A Study to Determine the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of ABBV-368 Plus Tilsotolimod and Other Therapy Combinations in Participants With Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Idera Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M19-894; 2019-003167-22 (EudraCT Number)
Record Dates: First submitted 2019-12-06; First posted 2019-12-12 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumors Cancer
Keywords: Squamous Cell Carcinoma; Head and Neck Squamous Cell Carcinoma; Locally Advanced Head and Neck Squamous Cell Carcinoma; Metastatic Head and Neck Squamous Cell Carcinoma; Cancer
MeSH Terms: conditions — Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck; Neoplasms | interventions — tilsotolimod; 130-nm albumin-bound paclitaxel; budigalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: ABBV-368 + Tilsotolimod (Experimental): Participants will be administered ABBV-368 and Tilsotolimod at various timepoints as described in the protocol.
  Interventions: Drug: ABBV-368; Drug: Tilsotolimod
- Arm 2: ABBV-368 + Tilsotolimod + Nab-paclitaxel (Experimental): Participants will be administered ABBV-368, Tilsotolimod and Nab-paclitaxel at various timepoints as described in the protocol.
  Interventions: Drug: ABBV-368; Drug: Tilsotolimod; Drug: Nab-paclitaxel
- Arm 3: ABBV-368 + Tilsotolimod + Nab-paclitaxel + ABBV-181 (Experimental): Participants will be administered ABBV-368, Tilsotolimod, Nab-paclitaxel and ABBV-181 at various timepoints as described in the protocol.
  Interventions: Drug: ABBV-368; Drug: Tilsotolimod; Drug: Nab-paclitaxel; Drug: ABBV-181

INTERVENTIONS:
Drug: ABBV-368 — Intravenous (IV) infusion
Drug: Tilsotolimod — Intratumoral (IT) injection
Drug: Nab-paclitaxel — Intravenous (IV) infusion
  Arms: Arm 2: ABBV-368 + Tilsotolimod + Nab-paclitaxel; Arm 3: ABBV-368 + Tilsotolimod + Nab-paclitaxel + ABBV-181
Drug: ABBV-181 — Intravenous (IV) infusion
  Other Names: Budigalimab
  Arms: Arm 3: ABBV-368 + Tilsotolimod + Nab-paclitaxel + ABBV-181

SUMMARY:
The main objective of this study is to assess safety, tolerability, and pharmacokinetics (PK) of ABBV-368 plus tilsotolimod; ABBV-368 plus tilsotolimod and nab-paclitaxel; and ABBV-368 plus tilsotolimod, nab-paclitaxel, and ABBV-181 in participants with recurrent/metastatic (R/M) head and neck squamous cell carcinoma (HNSCC).

ELIGIBILITY:
Inclusion Criteria:

* Participants should weigh at least 35 kg.
* Eastern Cooperative Oncology Group performance status of 0 or 1 and a life expectancy of >= 3 months.
* Participant have >= 1 lesion accessible for intratumoral injection.
* Histologically or cytologically confirmed R/M HNSCC (of the following 4 subsites: oral cavity, oropharynx, larynx, and hypopharynx) who previously progressed either during or after <= 3 prior treatment regimens administered in the recurrent or metastatic setting.

  * Must have received 1 immunotherapy regimen which included a PD-(L)1 inhibitor.
  * Must have received platinum-based therapy, or be considered ineligible for platinum-based therapy by the investigator.

Exclusion Criteria:

* Uncontrolled metastases to the central nervous system (CNS).

  * Participants with brain metastases are eligible provided that evidence of clinical and radiographic stable disease for at least 4 weeks after definitive therapy is given and participants have not used prohibited levels of steroids for at least 4 weeks prior to first dose of the study.
* Received prior treatment with OX40 or toll-like receptor (TLR) agonists (excluding topical agents).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to approximately 2 years following the first dose
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study.
Change in Vital Signs | Up to approximately 2 years following the first dose
  Number of participants with clinically significant change from baseline in vital signs like systolic and diastolic blood pressure will be reported.
Change in Clinical Laboratory Test Results | Up to approximately 2 years following the first dose
  Number of participants with clinically significant change from baseline in clinical laboratory test results like hematology will be reported.
Maximum Observed Serum Concentration (Cmax) of ABBV-368 | Cycle 1 through Cycle 3 (each cycle is approximately 28 days)
  Maximum Serum Concentration (Cmax) of ABBV-368
Time to Maximum Serum Concentration (Tmax) of ABBV-368 | Cycle 1 through Cycle 3 (each cycle is approximately 28 days)
  Time to Maximum Serum Concentration (Tmax) of ABBV-368
Area Under Serum Concentration-Time Curve of ABBV-368 From Time 0 to the Time of Last Measurable Concentration (AUCt) | Cycle 1 through Cycle 3 (each cycle is approximately 28 days)
  Area Under Serum Concentration-Time Curve of ABBV-368 From Time 0 to the Time of Last Measurable Concentration (AUCt)
Terminal-Phase Elimination Rate Constant (β) of ABBV-368 | Cycle 1 through Cycle 3 (each cycle is approximately 28 days)
  Terminal-Phase Elimination Rate Constant (β) of ABBV-368
Terminal Half-Life (t1/2) of ABBV-368 | Cycle 1 through Cycle 3 (each cycle is approximately 28 days)
  Terminal Half-Life (t1/2) of ABBV-368
Maximum Plasma Concentration (Cmax) of Tilsotolimod | Cycle 1 through Cycle 3 (each cycle is approximately 28 days)
  Maximum Observed Plasma Concentration (Cmax) of Tilsotolimod
Time to Maximum Plasma Concentration (Tmax) of Tilsotolimod | Cycle 1 through Cycle 3 (each cycle is approximately 28 days)
  Time to Maximum Plasma Concentration (Tmax) of Tilsotolimod
Area Under Plasma Concentration-Time Curve of Tilsotolimod From Time 0 to the Time of Last Measurable Concentration (AUCt) | Cycle 1 through Cycle 3 (each cycle is approximately 28 days)
  Area Under Plasma Concentration-Time Curve of Tilsotolimod From Time 0 to the Time of Last Measurable Concentration (AUCt)
Terminal-Phase Elimination Rate Constant (β) of Tilsotolimod | Cycle 1 through Cycle 3 (each cycle is approximately 28 days)
  Terminal-Phase Elimination Rate Constant (β) of Tilsotolimod
Terminal Half-Life (t1/2) of Tilsotolimod | Cycle 1 through Cycle 3 (each cycle is approximately 28 days)
  Terminal Half-Life (t1/2) of Tilsotolimod
Maximum Observed Serum Concentration (Cmax) of ABBV-181 (Arm 3 Only) | Cycle 1 through Cycle 3 (each cycle is approximately 28 days)
  Maximum Observed Serum Concentration (Cmax) of ABBV-181
Time to Maximum Serum Concentration (Tmax) of ABBV-181 (Arm 3 Only) | Cycle 1 through Cycle 3 (each cycle is approximately 28 days)
  Time to Maximum Serum Concentration (Tmax) of ABBV-181
Area Under Serum Concentration-Time Curve of ABBV-181 From Time 0 to the Time of Last Measurable Concentration (AUCt) (Arm 3 Only) | Cycle 1 through Cycle 3 (each cycle is approximately 28 days)
  Area Under Serum Concentration-Time Curve of ABBV-181 From Time 0 to the Time of Last Measurable Concentration (AUCt)
Terminal-Phase Elimination Rate Constant (β) of ABBV-181 (Arm 3 Only) | Cycle 1 through Cycle 3 (each cycle is approximately 28 days)
  Terminal-Phase Elimination Rate Constant (β) of ABBV-181
Terminal Half-Life (t1/2) of ABBV-181 (Arm 3 Only) | Cycle 1 through Cycle 3 (each cycle is approximately 28 days)
  Terminal Half-Life (t1/2) of ABBV-181

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 2 years following the first dose
  ORR is measured as the percentage of participants with a complete response (CR) or partial response (PR) as a confirmed response.
Clinical Benefit Rate (CBR) | Up to approximately 2 years following the first dose
  CBR is measured as the percentage of participants with a confirmed complete response (CR), confirmed partial response (PR), or stable disease (SD)
Time to Response (TTR) | Up to approximately 2 years following the first dose
  TTR is the time from date of first study drug exposure to the first instance of a complete response (CR) or partial response (PR) as a confirmed response, whichever occurs first.
Progression Free Survival (PFS) | Up to approximately 2 years following the first dose
  PFS is the time from date of first study drug exposure to disease progression or death, whichever occurs first.
Duration of Response (DOR) | Up to approximately 2 years following the first dose
  DOR is the time from the participant's initial response (CR or PR as a confirmed response) to disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (26):
- United States (8):
  - The University of Chicago Medical Center /ID# 217196, Chicago, Illinois
  - Norton Cancer Institute /ID# 216179, Louisville, Kentucky
  - Barbara Ann Karmanos Cancer In /ID# 214050, Detroit, Michigan
  - Nebraska Methodist Hospital /ID# 215786, Omaha, Nebraska
  - Atlantic Health System /ID# 216159, Morristown, New Jersey
  - Roswell Park Comprehensive Cancer Center /ID# 215882, Buffalo, New York
  - Vanderbilt Ingram Cancer Center /ID# 214040, Nashville, Tennessee
  - MD Anderson Cancer Center /ID# 214041, Houston, Texas
- France (4):
  - Centre Antoine Lacassagne - Nice /ID# 215706, Nice, Alpes-Maritimes
  - AP-HM - Hopital de la Timone /ID# 215657, Marseille, Bouches-du-Rhone
  - Hopital Saint-Andre /ID# 215702, Bordeaux, Gironde
  - Institut Curie /ID# 215653, Paris, Île-de-France Region
- Germany (3):
  - Universitaetsklinikum Erlangen /ID# 214196, Erlangen, Bavaria
  - Universitaetsklinikum Leipzig /ID# 214200, Leipzig, Saxony
  - Charite Universitaetsklinikum Berlin - Campus Benjamin Franklin /ID# 214197, Berlin
- Israel (3):
  - The Chaim Sheba Medical Center /ID# 215229, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus /ID# 215231, Haifa
  - Gastroenterology Institute, Division of Medicine /ID# 215862, Jerusalem
- Antoni van Leeuwenhoek /ID# 215291, Amsterdam, North Holland, Netherlands
- Spain (7):
  - Instituto Catalan de Oncologia (ICO) L'Hospitalet /ID# 221402, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Fuenlabrada /ID# 214263, Fuenlabrada, Madrid
  - Hospital Clinic de Barcelona /ID# 214264, Barcelona
  - Hospital Universitario 12 de Octubre /ID# 214198, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 214110, Madrid
  - Hospital Universitario Virgen de la Victoria /ID# 214109, Málaga
  - Hospital Clinico Universitario de Valencia /ID# 221401, Valencia

IPD SHARING:
Plan to Share IPD: No